CLINICAL TRIAL: NCT04870190
Title: To Evaluate the Efficacy and Safety of High-Dose Almonertinib Versus Osimertinib in the Second-Line Treatment of Patients With EGFR Mutations in Advanced NSCLC With Brain Metastases: a Multicenter, Randomized Controlled, Double-Blind Clinical Trial
Brief Title: Almonertinib Versus Osimertinib in the Patients With EGFR Mutations in Advanced NSCLC With Brain Metastases
Acronym: ATTACK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Chief physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YX-L-202106
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: NSCLC
MeSH Terms: interventions — aumolertinib; osimertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib (Experimental): Almonertinib will be administered orally at a dose of 165 mg per time, Q.D.
  Interventions: Drug: Almonertinib
- Osimertinib (Active Comparator): Osimertinib will be administered orally at a dose of 80 mg per time, Q.D.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib will be administered orally at a dose of 165 mg per time, Q.D.
  Other Names: HS-10296
  Arms: Almonertinib
Drug: Osimertinib — Osimertinib will be administered orally at a dose of 80 mg per time, Q.D.
  Other Names: Teresa; AZD9291
  Arms: Osimertinib

SUMMARY:
This is a multicenter, randomized controlled, double-blind clinical trial. The study is designed to evaluate the efficacy and safety of high-dose Almonertinib versus Osimertinib in the second-line treatment of patients with EGFR mutations in advanced NSCLC with brain metastases.

DETAILED DESCRIPTION:
This is a multicenter, randomized controlled, double-blind clinical study which will recruit about 232 patients in China.

The study is designed to evaluate the efficacy and safety of high-dose Almonertinib versus Osimertinib in the second-line treatment of patients with EGFR mutations in advanced NSCLC with brain metastases.

Target Patient Population:Age 18 years or older with histologically or cytologically proven advanced NSCLC with brain parenchymal (BM) metastases.The patient was laboratory confirmed to be EGFR T790M mutation positive at or after progression of 1/2 generation EGFR-TKI therapy.

Test Drug, Dosage and Medication Regimen:Almonertinib will be administered orally at a dose of 165 mg per time, Q.D.If a patient cannot tolerate a dose of 165mg due to adverse reactions, when the adverse reactions restore to level 1 (CTCAE 5.0) or below, the dosage could be adjusted to 110mg per day, Q.D.

Osimertinib will be administered orally at a dose of 80 mg per time, Q.D. If a patient cannot tolerate a dose of 40mg due to adverse reactions, when the adverse reactions restore to level 1 (CTCAE 5.0) or below, the dosage could be adjusted to 40mg per day, Q.D.

ELIGIBILITY:
Inclusion Criteria:

1.18 ≤ age and above. 2. Histology or cytology is confirmed as NSCLC, imaging confirmed as advanced NSCLC with brain metastasis (including relapsed or newly diagnosed advanced patients after previous surgical treatment; according to AJCC eighth edition lung cancer staging standard).

3. Progressed after receiving first or second generation EGFR-TKI treatment, T790M positive.

4. According to RECIST1.1, the patient has at least 1 intracranial target lesion and 1 extracranial target lesion. The requirements for target lesions are: measurable lesions that have not undergone local treatment such as irradiation or have clearly progressed after local treatment, with the longest diameter at baseline ≥10 mm (if it is a lymph node, the maximum short diameter is required to be ≥15 mm).

5. The brain condition is stable for at least 2 weeks before the study drug treatment, without any systemic (oral or parenteral) corticosteroid or anticonvulsant drug treatment. Non-absorbable corticosteroids can be used locally and inhaled according to the indications.

6. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0 or 1, and there is no deterioration at least 2 weeks before the study drug treatment, and the expected survival period is not less than 12 weeks.

7. Female patients of childbearing age are willing to take appropriate contraceptive measures from signing the informed consent to 6 months after the last treatment with the study drug and should not breastfeed; male patients are willing from signing the informed consent to 6 months after the last treatment with the study drug Use barrier contraception (ie condoms).

8. Female patients of childbearing age must have a negative serum or urine HCG test within 7 days before enrollment in the study, and they must be non-lactating.

9.The subjects themselves participated voluntarily and signed a written informed consent form.

Exclusion Criteria:

1. Have received any of the following treatments:

   1. Within 4 weeks before the first administration of the study drug, the patient has undergone major surgery (such as craniotomy, thoracotomy, or laparotomy, etc.), or underwent minor traumatic surgery (biopsy, bronchoscopy, and Thoracic drainage). The definition of major surgery refers to the level 3 and level 4 surgery specified in the "Administrative Measures for the Clinical Application of Medical Technology" in Appendix H, which was implemented on November 1, 2018;
   2. Except for patients who have received local radiotherapy (palliative radiotherapy for bone in non-target lesions) within 2 weeks before the first administration of the study drug; within 4 weeks before the first administration of the study drug, they have received more than 30% bone marrow irradiation (calculated area of bone marrow) See Annex I), or received extensive radiotherapy; received whole brain radiotherapy due to this disease before enrollment;
   3. Recurrence within 6 months after adjuvant or neoadjuvant treatment for early lung cancer; if there is both neoadjuvant therapy and adjuvant therapy, the adjuvant treatment time will be calculated;
   4. There is pleural effusion/peritoneal effusion that requires clinical intervention (patients who do not need to drain the effusion or who are stable for 2 weeks or more after drainage can be included); there is pericardial effusion (a small amount of pericardium that is stable for 2 weeks or more) Fluid effusion is allowed to enter the group). If anti-tumor drugs have been used locally (such as chest cavity perfusion) during drainage, at least 5 drug half-lives or 21 days (whichever is shorter) must be eluted before the first administration of the study treatment before being included in the group;
   5. Within 7 days before the first administration of the study drug, have used CYP3A4 strong inhibitors, strong inducers or drugs with a narrow therapeutic window of sensitive substrates, or need to continue to receive these drugs during the study period (see Appendix E for the list of drugs);
   6. Are receiving drugs that are known to prolong the QT interval or may cause torsades de pointes, or need to continue to receive these drugs during the study period (see Appendix E for the drug list and washout time);
   7. Within 4 weeks before the first administration of the study drug, the five half-lives of the study drug as a subject participating in other clinical trials or still in other clinical trials, whichever is longer (except for screening failure).
2. Mixed SCLC and mixed NSCLC, large cell neuroendocrine carcinoma and sarcomatoid carcinoma confirmed by histology or cytology.
3. At the beginning of the study drug treatment, there is a residual toxicity of the previous anti-tumor treatment that is greater than CTCAE level 1 that has not been relieved, except for hair loss and level 2 neurotoxicity caused by the previous anti-tumor. In the past, intracranial hemorrhage unrelated to the tumor occurred.
4. History of other primary malignant tumors, except for the following:

   1. Malignant tumors that have been cured, have been inactive for ≥ 5 years and have a very low risk of recurrence before being selected for the study;
   2. Non-melanoma skin cancer or malignant freckle-like nevus that has been adequately treated and has no evidence of disease recurrence;
   3. Carcinoma in situ with adequate treatment and no evidence of disease recurrence.
5. Diagnosis of meningeal metastasis by clinical symptoms or imaging or cerebrospinal fluid, or brain parenchymal metastasis combined with meningeal metastasis.
6. Patients who are allergic to MRI contrast agent gadolinium or who cannot tolerate MRI examinations (such as pacemakers, metals in the body, etc.).
7. Any serious or poorly controlled systemic disease, as determined by the investigator, such as poorly controlled hypertension, active bleeding susceptibility, or active infection. There is no need to screen for chronic diseases.
8. Clinically serious abnormal gastrointestinal function, which may affect the intake, transport or absorption of drugs, such as inability to take drugs, uncontrollable nausea or vomiting, history of extensive gastrointestinal resection, uncured recurrent diarrhea, atrophy Gastritis, uncured gastric diseases that require proton pump inhibitors for a long time, Crohn's disease, ulcerative colitis, etc.
9. Hepatic encephalopathy, hepatorenal syndrome or cirrhosis.
10. Meet any of the following cardiac examination results:

    1. The average QT interval (QTcF) corrected by Fridericia's formula obtained from 3 ECG examinations in the resting state> 470 msec;
    2. Resting ECG prompts the existence of various clinically significant rhythms, conduction or ECG morphological abnormalities judged by the investigator (such as complete left bundle branch block, 3 degree atrioventricular block, 2 degree atrium Ventricular block and PR interval> 250 msec, etc.);
    3. There are any factors that increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death or prolonged QT of immediate family members under the age of 40 Any concomitant drugs in the interval;
    4. Left ventricular ejection fraction (LVEF) <50%.
11. Insufficient bone marrow reserve or organ function, reaching any of the following laboratory limits (no corrective treatment within 1 week before laboratory examination of blood):

    1. Absolute neutrophil count <1.5×109/L;
    2. Platelet count<100×109/L;
    3. Hemoglobin <90 g/L (<9 g/dL);
    4. If there is no clear liver metastasis, alanine aminotransferase> 2.5 times the upper limit of normal (ULN); if there is liver metastasis, alanine aminotransferase> 5×ULN;
    5. If there is no clear liver transfer, aspartate aminotransferase> 2.5×ULN; if there is liver transfer, aspartate aminotransferase> 5×ULN;
    6. If there is no clear liver metastasis, total bilirubin> 1.5×ULN; or Gilbert syndrome (unconjugated hyperbilirubinemia) or liver metastasis, total bilirubin> 3×ULN;
    7. Creatinine>1.5×ULN and creatinine clearance rate<50 mL/min (calculated by Cockcroft-Gault formula); only when creatinine>1.5×ULN, creatinine clearance rate needs to be confirmed;
    8. Serum albumin (ALB) <28 g/L;
12. Infections in which pathogenic bacteria that are currently producing symptoms or diseases that require systemic treatment are rapidly multiplying, that is, active infections. Including active fungal, bacterial and/or viral infections (such as HBV, HIV, etc.).
13. Female subjects who are pregnant, lactating, or planning to become pregnant during the study period.
14. A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
15. Have a history of hypersensitivity to any active or inactive ingredients of Almonertinib or to drugs with similar chemical structure or the same class of Almonertinib.
16. Any serious or uncontrolled eye disease (especially severe dry eye syndrome, dry keratoconjunctivitis, severe exposure keratitis or other diseases that may increase epithelial damage) may increase the safety of patients by the doctor's judgment Sexual risk.
17. Patients who may have poor compliance with the research procedures and requirements, such as patients who have a clear history of neurological or psychiatric disorders (including epilepsy or dementia), and currently suffer from mental disorders, etc., as judged by the investigator.
18. The investigator judges that there are any patients with conditions that endanger the safety of the patient or interfere with the evaluation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival (IPFS) in patients with advanced NSCLC with brain metastases treated with high-dose Almonertinib versus Osimertinib in second-line treatment with positive EGFR T790M mutation. | 36 months
  To evaluate the efficacy of high dose Almonertinib versus Osimertinib by IRC(RECIST 1.1).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 36 months
  To evaluate the safety of high dose Almonertinib versus Osimertinib.

IPD SHARING:
Plan to Share IPD: No